CLINICAL TRIAL: NCT06521567
Title: Phase 1/2 Dose Determination and Dose Expansion Study of Cobolimab in Combination With Dostarlimab in Pediatric and Young Adult Participants With Newly Diagnosed and Relapsed/Refractory Tumors (POPSTAR)
Brief Title: A Study of Cobolimab Plus Dostarlimab in Pediatric and Young Adult Participants With Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 219451; 2024-511350-41-00 (Other: EU CT Number)
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Melanoma; Hodgkin Lymphoma; High and Low Grade Glioma; Glioblastoma Multiforme (GBM); Diffuse Intrinsic Pontine Glioma (DIPG); Ependymoma; Osteosarcoma; Hepatic Tumors; Hepatoblastoma; Hepatocellular Carcinoma (HCC); Fibrolamellar Carcinoma; Rhabdomyosarcoma
Keywords: Solid Tumours; Cobolimab; Dostarlimab
MeSH Terms: conditions — Melanoma; Hodgkin Disease; Glioblastoma; Diffuse Intrinsic Pontine Glioma; Ependymoma; Osteosarcoma; Carcinoma, Hepatocellular; Hepatoblastoma; Fibrolamellar hepatocellular carcinoma; Rhabdomyosarcoma | interventions — dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1- Dose determination (Experimental)
  Interventions: Drug: Cobolimab; Drug: Dostarlimab
- Part 2- Dose expansion (Experimental)
  Interventions: Drug: Cobolimab; Drug: Dostarlimab

INTERVENTIONS:
Drug: Cobolimab — Cobolimab will be administered
Drug: Dostarlimab — Dostarlimab will be administered

SUMMARY:
The goal of this interventional study is to determine the strength of cobolimab and dostarlimab that is most tolerated in children and young adults who have advanced solid tumors. This study also aims: (a) to check if it is safe to use cobolimab and dostarlimab combination in children and young adults, (b) to see how to manage the side effects that may occur, and (c) the effect of this treatment in participants

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Participants between the age of 0 to not more than 21 years at the time of signing informed consent form (ICF).
* Disease characteristics:

Part 1: Participants with advanced or metastatic solid tumors who have had disease progression after treatment with available therapies that are known to confer clinical benefit and who have limited available treatment options as determined by the investigator. Additionally, exposure to prior immunotherapy or experimental therapies is acceptable:

1. Melanoma
2. Hodgkin Lymphoma
3. High and Low Grade Glioma: including Glioblastoma multiforme (GBM), Diffuse intrinsic pontine glioma (DIPG), and ependymoma.
4. Osteosarcoma
5. Hepatic tumors [including Hepatoblastoma, Hepatocellular carcinoma (HCC), and Fibrolamellar carcinoma]
6. Rhabdomyosarcoma

Part 2:

1. Participants with Melanoma who have not received prior systemic therapy:

   * Participants with BRAF gene, found on chromosome 7 (BRAF) mutations who are eligible for a BRAF-targeted therapy are eligible if they qualify for immunotherapy.
   * Participants with locally treated and controlled metastatic central nervous system (CNS) lesions without leptomeningeal spread are eligible
2. Relapsed/refractory Hodgkin lymphoma (HL) that has failed at least 2 prior lines of systemic therapy)

   * Participants must have performance status >=60 percent (%) on the Karnofsky scale for participants >16 years of age and >=60% on the Lansky scale for participants <=16 years of age.
   * Adequate organ function as demonstrated by a complete blood count at screening obtained without transfusion [platelets or red blood cells (RBC)] or receipt of Colony stimulating factor (CSF), Granulocyte colony stimulating factor (G-CSF), Granulocyte macrophage colony stimulating factor (GMCSF) or rErythropoeitin (rEPO) within 2 weeks prior to screening.
   * Adolescent participants who have entered puberty must consent (be willing) to use of contraceptive measures, or refrain from sexual intercourse, if in line with their usual practice, as well as sperm/egg donation for the duration of treatment

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical conditions:

* Participant has uncontrolled CNS involvement by any tumor pathology
* Participant has a heart rate-corrected QT interval according to QT interval (corrected) (Friderecia's formula) (QTcF) prolongation at screening >470 millisecond (msec) or >480 msec for participants with bundle branch block.
* Participant has clinically significant cardiovascular disease
* Participant has chronic respiratory disease
* Participant has known sensitivity to study intervention components or excipients or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Participants who have a history of immunodeficiency disease, including other acquired or congenital immunodeficiency diseases, or organ transplantation
* Participants who have received plasma exchange within 7 days before the first dose of study intervention.
* Participant has current active pneumonitis or any history of pneumonitis requiring steroids or immunomodulatory treatment within 90 days of planned enrollment or any history of drug-induced pneumonitis.
* Participant has a history of autoimmune disease that has required systemic treatments in the 2 years prior to screening. Participants with prior history of autoimmune disease must be discussed with the medical monitor. Replacement therapy is not considered a form of systemic therapy (e.g., thyroid hormone for autoimmune thyroiditis or insulin is not exclusionary)
* Participant has ongoing adverse reaction(s) from prior therapy that has (have) not recovered to ≤Grade 1 or to the Baseline status preceding prior therapy, excluding [e.g., alopecia, hearing loss, vitiligo, endocrinopathy managed with replacement therapy, and Grade 2 neuropathy], or that the investigator, with the agreement of the sponsor, considers to be not clinically relevant for the tolerability of study intervention in the current clinical study.
* Participant has any active renal condition (e.g., infection, requirement for dialysis, or any other significant renal condition (that could affect the participant's safety).
* Participant has any serious and/or unstable medical or psychiatric disorder or other condition(s) (including laboratory assessment abnormalities) that could interfere with the participant's safety, obtainment of informed consent, or compliance to the study procedures.

Prior/ Concomitant therapy:

* Has received treatment with an investigational agent or any other anti-cancer therapy within 30 days, or <5 times the half-life of the most recent therapy prior to signing ICF, whichever is shorter.
* Has received systemic steroid therapy within 3 days prior to the first dose of the study treatment or is receiving any other form of immunosuppressive medication. Replacement therapy is not considered a form of systemic therapy. Use of inhaled corticosteroids, local steroid injection, or steroid eye drops is allowed.
* Has not met the following waiting/washout periods for X-ray therapy (XRT) including external beam radiation therapy/external beam irradiation including protons:
* Participant has had major surgery within 28 days prior to the first dose of study treatment or has not adequately recovered from any AEs (Grade ≤1) and/or complications from any major surgery. Surgical implantation of a port catheter is not exclusionary.
* Prior Bone Marrow Transplant <60 days of screening.
* Participant has experienced Grade 3 or higher hypersensitivity to prior monoclonal antibody therapy.

Prior/Concurrent clinical study experience

* Is currently enrolled or has participated in any other clinical study involving an investigational study or interventional medical research within 21 days or 5 half-lives, whichever is shorter, of an investigational medicinal product before signing ICF Diagnostic assessments
* Has documented presence of Hepatitis B surface antigen (HbsAg) at Screening or within 3 months prior to first dose of study intervention.
* Has a positive Hepatitis C virus (HCV) antibody test result at Screening or within 3 months prior to first dose of study intervention.
* Has a positive HCV Ribonucleic Acid (RNA) test result at Screening or within 3 months prior to first dose of study intervention.
* Has a known history of Human immunodeficiency virus (HIV) or has a HIV-positive test result at Screening.
* Is pregnant or breastfeeding.

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-10-13 (Estimated); Study Completion 2026-10-13 (Estimated)

PRIMARY OUTCOMES:
Part 1- Number of participants with Dose Limiting Toxicities (DLTs) | Up to 42 days
Part 1- Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), immune-mediated adverse events (imAEs) and adverse events (AEs) leading to discontinuation occurring during the study | Up to approximately 46 months
Part 1- Serum concentration of Cobolimab | 1±0.5 hours (h) post-dose on Cycle 1 Day 1; 168±12 h post-dose Cycle 1Day 8; Pre-dose and 1±0.5 h post-dose on Cycle 2 Day 1; Cycle 4 Day 1 and Cycle 6 Day 1(Each cycle is of 21 days)
Part 1- Serum concentration of Dostarlimab | 1±0.5 h post start of cobolimab infusion on Cycle 1 Day 1; Pre-dose on Cycle 2 Day 1; Cycle 4 Day 1 and Cycle 6 Day 1(Each cycle is of 21 days)
Part 1- Recommended Phase 2 Dose (RP2D) of Cobolimab and Dostarlimab combination | Up to approximately 12 months
Part 2- Confirmed Objective Response Rate (ORR) | Up to approximately 46 months
  Confirmed ORR is defined as the proportion of participants who have achieved confirmed complete response (CR) or confirmed partial response (PR), evaluated using disease-specific tumor assessment criteria based on Investigator assessment
Part 2- Number of participants with TEAEs, SAEs, imAEs, TEAEs leading to death and AEs leading to discontinuation | Up to approximately 46 months
Part 2-Number of participants with changes in laboratory parameters, vital signs and cardiac parameters | Up to approximately 46 months

SECONDARY OUTCOMES:
Part 1 and 2: Receptor occupancy (RO) | Pre-dose Cycle 1 Day 1, 5 h post-start of cobolimab administration Cycle 1 Day 1, anytime Cycle 1 Day 8, pre-dose Cycle 2 Day 1, and pre-dose Cycle 4 Day 1 (Each cycle is of 21 days)
  RO will be measured in whole blood and presented as normalized ratio [Fluorescence Minus One (FMO) subtracted values of free T cell immunoglobulin and mucin domain containing protein 3 (TIM-3) to total TIM-3]
Part 1- Confirmed ORR | Up to approximately 70 months
  Confirmed ORR is defined as the proportion of participants who have achieved confirmed CR or confirmed PR, evaluated using disease specific tumor assessment criteria based on Investigator assessment
Part 1 and 2: Progression Free Survival (PFS) | Up to approximately 70 months
  PFS is defined as the length of time until disease progression, from the date of first dose to the earliest date of assessment of disease progression based on disease-specific tumor assessment criteria by Investigator assessment, or death by any cause, whichever occurs first
Part 1 and 2: Duration of response (DOR) | Up to approximately 70 months
  DOR is defined as the time from first documented response (CR/PR) until the time of first documentation of disease progression based on disease-specific tumor assessment criteria by Investigator assessment, or death, whichever occurs first
Part 1 and 2: Overall Survival (OS) | Up to approximately 70 months
  OS is defined as the time from the date of first dose to the date of death by any cause
Part 1 and 2: Number of participants with positive results in Anti-drug antibody (ADA) test against Cobolimab | Pre-dose on Cycle 1 Day 1; Cycle 2 Day 1; Cycle 4 Day 1 and Cycle 6 Day 1[Each cycle is of 21 days]; 30-Day and 90-Day safety follow up (FUP) Visit
Part 1 and 2: Number of participants with positive results in Anti-drug antibody (ADA) test against Dostarlimab | Pre-dose on Cycle 1 Day 1; Cycle 2 Day 1; Cycle 4 Day 1 and Cycle 6 Day 1[Each cycle is of 21 days]; 30-Day and 90-Day safety follow up (FUP) Visit
Part 1 and 2: Titers of ADA to Cobolimab | Pre-dose on Cycle 1 Day 1; Cycle 2 Day 1; Cycle 4 Day 1 and Cycle 6 Day 1[Each cycle is of 21 days]; 30-Day and 90-Day safety follow up (FUP) Visit
Part 1 and 2: Titers of ADA to Dostarlimab | Pre-dose on Cycle 1 Day 1; Cycle 2 Day 1; Cycle 4 Day 1 and Cycle 6 Day 1[Each cycle is of 21 days]; 30-Day and 90-Day safety follow up (FUP) Visit
Part 2- Serum concentration of Cobolimab | 1±0.5 hours(h) post-dose on Cycle1Day 1;168±12h post-dose Cycle1Day8; Pre-dose & 1±0.5h post-dose on Cycle2Day1; Cycle4Day1 & Cycle6Day1[Each cycle is of 21 days];End of Treatment(EOT; EOT is within 7days of last dose), 30Day safety follow up(FUP) Visit
Part 2- Serum concentration of Dostarlimab | 1±0.5 h post start of cobolimab infusion on Cycle 1 Day 1; Pre-dose on Cycle 2 Day 1; Cycle 4 Day 1 and Cycle 6 Day 1 [Each cycle is of 21 days]; End of Treatment (EOT; EOT is within 7 days of last dose), 30-Day safety follow up (FUP) Visit

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (19):
- United States (6):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Hackensack, New Jersey
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Madison, Wisconsin
- Czechia (2):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Phaha 5
- GSK Investigational Site, Copenhagen, Denmark
- France (5):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Villejuif
- Italy (2):
  - GSK Investigational Site, Bologna
  - GSK Investigational Site, Napoli
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/